CLINICAL TRIAL: NCT01268371
Title: Comparison of Biolimus-eluting Biodegradable Polymer, Everolimus-eluting and Sirolimus-eluting Coronary Stents
Acronym: BESS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Seung-Jea Tahk, Dr., Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BESS
Record Dates: First submitted 2010-12-29; First posted 2010-12-30 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Promus Element (Active Comparator): Everolimus-eluting stent
  Interventions: Device: Promus Element, Boston Scientific Corporation
- Nobori (Active Comparator): Biolimus-eluting stent with biodegradable polymer
  Interventions: Device: Nobori, Terumo Corporation (Japan)

INTERVENTIONS:
Device: Promus Element, Boston Scientific Corporation — Everolimus-eluting stent
  Other Names: Everolimus-eluting stent
  Arms: Promus Element
Device: Nobori, Terumo Corporation (Japan) — Biolimus-eluting stent with biodegradable polymer
  Other Names: Biolimus-eluting stent with biodegradable polymer
  Arms: Nobori

SUMMARY:
To compare the safety and efficacy of coronary stenting with everolimus-eluting stent (Promus Element®) and biolimus-eluting stent with biodegradable polymer (Nobori®)

ELIGIBILITY:
Inclusion Criteria:

* Significant coronary artery stenosis (> 50% by visual estimate)
* Stable angina, unstable angina, Non-ST elevation myocardial infarction (NSTEMI) and documented silent ischemia
* Patients eligible for intracoronary stenting
* age ≥ 20 years old

Exclusion Criteria:

* ST segment elevation myocardial infarction (within 24 hours)
* Low ejection fraction (< 25%)
* Cardiogenic shock
* History of bleeding diathesis or known coagulopathy
* Limited life-expectancy (less than 1 year) due to combined serious disease
* Contraindication to heparin, sirolimus, everolimus and biolimus
* Contraindication to aspirin and clopidogrel
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1462 (Estimated)
Dates: Start 2010-12; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The Number of Participants with Majour Adverse Cardiac Events (composite of death, myocardial infarction, target vessel revascularization and stent thrombosis | 1 year after index procedure

SECONDARY OUTCOMES:
The number of participants with majour adverse cardiac events (composite of death, myocardial infarction, target vessel revascularization and stent thrombosis | 2 years after index procedure
Death (all-cause and cardiac) | 1 to 2 years after index procedure
Myocardial infarction (Q wave and non-Q wave) | 1 to 2 years after index procedure
Target vessel revascularization (ischemia- and clinically-driven) | 1 to 2 years after index procedure
Target lesion revascularization (ischemia- and clinically-driven) | 1 to 2 years after index procedure
Stent thrombosis | 1 to 2 years after index procedure
In-stent and in-segment late loss at 1 year angiographic follow-up | 1 year after index procedure
In-stent and in-segment restenosis at 1 year angiographic follow-up | 1 year after index procedure
Incidence and angiographic pattern of restenosis at 1 year angiographic follow-up | 1 year after index procedure
The incidence of Procedural success | index procedure (day 0)
The number of participants with death and myocardial infarction | 1 to 2 years after index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jea Tahk, MD, PhD, Principal Investigator — Department of Cardiology, Ajou University School of Medicine
Locations (26):
- South Korea (26):
  - Hallym University Sacred Heart Hospital, Anyang
  - Sejong Hospital, Bucheon-si
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Kangwon National University Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Konyang University Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Inje University ilsan Paik Hospital, Ilsan
  - Gachon University Gil Hospital, Incheon
  - Cheju Halla General Hospital, Jeju City
  - Pusan National University Hospital, Pusan
  - Hallym University Hankang Sacred Heart Hospital, Seoul
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Kyunghee University Medical Center, Seoul
  - The Catholic University of Korea Seoul ST. Mary's Hospital, Seoul
  - Yonsei University Gangnam Severance Hospital, Seoul
  - St. Carollo Hospital, Suncheon
  - Ajou University Medical Center, Suwon
  - Catholic University ST. Vincent's Hospital, Suwon
  - Ulsan University Hospital, Ulsan
  - Yonsei University Wonju College of Medicine Wonju Christion Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan